CLINICAL TRIAL: NCT07338838
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of TQB3142 for Injection in Patients With Advanced Malignant Tumors
Brief Title: To Evaluate the Tolerability and Pharmacokinetics of TQB3142 for Injection in Patients With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3142-I-01
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3142 injection (Experimental): The drug was administered every weeks for 28 consecutive days in a treatment cycle.
  Interventions: Drug: TQB3142 injection

INTERVENTIONS:
Drug: TQB3142 injection — TQB3142 for injection is a B-cell lymphoma-extra large inhibitor.

SUMMARY:
To explore the safety, tolerability and pharmacokinetics of TQB3142 for injection in subjects with advanced malignant tumors

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and had good compliance;
* 18 years old ≤ age ≤75 years old (calculated on the date of signing the informed consent);
* Eastern Cooperative Oncology Group Performance Status (ECOG) score 0~1;
* Expected survival greater than 12 weeks;
* Patients with advanced tumors confirmed by cytology/histopathology, failure of standard treatment or lack of effective treatment;
* Evidence of at least one measurable lesion according to RECIST 1.1 criteria；
* The main organs function well and meet the following criteria:

  1. Hemoglobin (HGB) ≥90g/L;
  2. Absolute neutrophil count (ANC) of solid tumor subjects ≥1.5×109 /L;
  3. Platelet count (PLT) ≥100×109/L；
  4. Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN);
  5. Alanine transferase (ALT) and aspartate transferase (AST) ≤2.5×ULN. ALT and AST≤5×ULN if accompanied by liver metastasis;
  6. Serum creatinine (CR) ≤1.5×ULN or creatinine clearance (CCR) ≥60 mL /min (standard Cockcroft-Gault formula was applied;
  7. Prothrombin time (PT), activated partial thromboplastin time (APTT), International standardized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy);
* Women of reproductive age should agree that effective contraception must be used during the study period and for 6 months after the end of the study, and that serum or urine pregnancy tests are negative within 7 days prior to study enrollment; Men should agree that effective birth control must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

I. Comorbid Conditions and Medical History:

* Any active malignancy within the 3 years prior to the first dose, except for the specific cancer under study in this trial and locally recurrent cancers that have been cured (e.g., resected basal cell or squamous cell skin cancer, superficial bladder cancer [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the lamina propria)], carcinoma in situ of the cervix, or carcinoma in situ of the breast).
* Failure to recover from toxicities and/or complications of prior interventions to ≤ Grade 1 per CTCAE, except for alopecia and peripheral neuropathy ≤ Grade 2.
* Receipt of any blood product transfusion or requirement for hematopoietic growth factor therapy within 28 days prior to the first dose.
* Bleeding Risk:

  1. Known bleeding diathesis or disorder.
  2. History of non-chemotherapy-induced thrombocytopenic bleeding or history of platelet transfusion refractoriness within 1 year prior to the first dose.
  3. Presence or high suspicion of active bleeding/hemolytic disorders such as Immune Thrombocytopenic Purpura (ITP), Autoimmune Hemolytic Anemia (AIHA), Evans Syndrome, Hemolytic Uremic Syndrome, Thrombotic Thrombocytopenic Purpura (TTP), Disseminated Intravascular Coagulation (DIC).
  4. Requirement for warfarin, aspirin, or other anticoagulant/antiplatelet agents for any reason within 28 days prior to treatment initiation.
  5. Uncontrolled or CTCAE ≥ Grade 2 bleeding events (e.g., gastrointestinal bleeding) or history of hemoptysis (> 2.5 mL of fresh blood per day) within 90 days prior to the first dose.
  6. Major surgical treatment or significant traumatic injury (excluding procedures like needle biopsy, endoscopic biopsy) within 28 days prior to the first dose.
  7. Non-healing wounds or fractures (excluding pathological fractures).
* Arterial/venous thrombotic events within 6 months prior to the first dose, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
* History of drug (psychoactive substances) or alcohol abuse with inability to abstain, or presence of psychiatric disorders.
* Subjects with any severe and/or uncontrolled diseases, including:

  1. Poorly controlled blood pressure (systolic BP ≥ 150 mmHg or diastolic BP ≥ 100 mmHg) despite treatment with two or more antihypertensive medications.
  2. Myocardial ischemia or myocardial infarction ≥ Grade 2, arrhythmias, and congestive heart failure ≥ Grade 2 (NYHA classification).
  3. History or presence of non-infectious pneumonitis requiring corticosteroid treatment (including but not limited to Acute Respiratory Distress Syndrome, Acute Hypersensitivity Pneumonitis, Drug-Related Pneumonitis, Bronchospasm, Acute Interstitial Pneumonia, Idiopathic Pulmonary Fibrosis, etc.).
  4. History, presence, or suspicion of Chronic Obstructive Pulmonary Disease (COPD) with Forced Expiratory Volume in 1 second (FEV1) < 60% of predicted value.
  5. Active or uncontrolled severe infection (≥ CTCAE Grade 2 infection).
  6. Diagnosis of Coronavirus Disease 2019 (COVID-19) infection within 3 months prior to the first dose.
  7. Decompensated cirrhosis (Child-Pugh class B or C), active hepatitis:

     * Hepatitis B reference: Hepatitis B Virus (HBV) - DNA > 1*10³ copies/mL or >2000 IU/mL if HBsAg positive.
     * Hepatitis C reference: Hepatitis C Virus (HCV) RNA above the upper limit of normal.

     (Note: Eligible subjects who are HBsAg positive or anti-Hepatitis B core (HBc) antigen positive, or have hepatitis C, require continuous antiviral therapy to prevent viral reactivation.)
  8. Active syphilis.
  9. Renal abnormalities:

     * Renal failure requiring hemodialysis or peritoneal dialysis.
     * History or presence of nephrotic syndrome (except if cured), chronic nephritis.
  10. History of immunodeficiency, including HIV positivity or other acquired/congenital immunodeficiency diseases; history of active autoimmune disease or autoimmune diseases including but not limited to Crohn's disease, ulcerative colitis, autoimmune hepatitis/enteritis/vasculitis/nephritis, etc.; or history of organ transplantation (except corneal transplant).
  11. Presence or history of autoimmune disease requiring treatment. Subjects with hypothyroidism on stable replacement therapy or Type 1 diabetes mellitus may be eligible.
  12. Urinalysis showing urine protein ≥ ++, and confirmed 24-hour urinary protein > 1.0 g (except for subjects with multiple myeloma).
  13. Poorly controlled diabetes (Fasting Blood Glucose > 10 mmol/L).
  14. Epilepsy requiring treatment.

II. Tumor-Related Symptoms and Treatment:

* Known central nervous system (CNS) involvement or carcinomatous meningitis; subjects with solid tumors who have received treatment for brain metastases and have been clinically stable for at least 28 days prior to the first dose without requiring steroids or other therapy for brain metastases may be eligible.
* Prior chemotherapy, targeted therapy, radiotherapy, or other anti-tumor therapy within 4 weeks before the first dose (calculation based on the end date of the last treatment for washout period).
* Prior allogeneic hematopoietic stem cell transplantation, autologous hematopoietic stem cell transplantation, or other cell therapies (e.g., Chimeric Antigen Receptor T-cell [Chimeric Antigen Receptor T-cell Therapy (CAR-T)] therapy).
* Treatment within 2 weeks prior to the first dose with Chinese patent medicines approved by the National Medical Products Administration (NMPA) with clearly stated anti-tumor indications in their package inserts (including Fufang Banmao Capsule, Kang'ai Injection, Kanglaite Capsule/Injection, Aidi Injection, Yadanzi Oil Injection/Capsule, Xiaoaiping Tablet/Injection, Huachansu Capsule, etc.).
* Serous cavity (pleural, peritoneal, or pericardial) effusion requiring repeated drainage for symptomatic relief (investigator's judgment), or receipt of therapeutic serous cavity effusion drainage within 2 weeks prior to treatment.
* Imaging (CT or MRI) showing tumor invasion of major blood vessels, or the investigator judges a high probability of fatal hemorrhage due to tumor invasion of major blood vessels during the study period.

III. Study Treatment-Related:

* Prior treatment with B-cell lymphoma-extra large (Bcl-xL) inhibitors.
* History of live attenuated vaccination within 4 weeks prior to the first dose or planned live attenuated vaccination during the study period.
* Known allergy to any component of the study drug(s).
* Requirement for or use of strong inhibitors or inducers of Cytochrome P450 3A (CYP3A) within 2 weeks prior to the first dose (medications or food).
* Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered systemic treatment.
* Diagnosis of immunodeficiency or current systemic glucocorticoid therapy (at a dose equivalent to >10 mg/day prednisone or equivalent) or any other form of immunosuppressive therapy (including but not limited to cyclosporine A, tacrolimus, cyclophosphamide, etc.) continued within 2 weeks prior to study treatment initiation. Exceptions include: ① Topical, ocular, intra-articular, intranasal, or inhaled corticosteroids are permitted. ② Short-term use of corticosteroids for prophylaxis (e.g., contrast allergy) or treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction from contact allergen) is permitted.
* Participation in another anti-tumor drug clinical trial within 4 weeks prior to the first dose or within 5 drug half-lives (whichever is shorter).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Phase II recommended doses (RP2D) | Up to 24 months
  The dosage of drug therapy recommended for use in the second phase of clinical trials (i.e., phase II clinical trials).
Dose-limiting toxicity (DLT) | Up to 1 month
  Adverse events that meet the protocol definition of dose-limiting toxic event timing were evaluated according to the Common Terminology Criteria for Adverse Events 5.0.
Maximum tolerated dose (MTD) | Up to 1 month
  The previous dose of the dose group in which dose-limiting toxicity occurs is the maximum tolerated dose.

SECONDARY OUTCOMES:
Numbers of participant with incidence and severity of Adverse Event (AE) and Serious Adverse Event (SAE), and abnormal laboratory test indicators | Up to 24 months
  Numbers of participant with incidence and severity of AE and SAE, and abnormal laboratory test indicators.
Peak time | Up to 4 month
  Time to peak blood concentration after a single dose
Objective response rate | Up to 24 months
  The objective response rate of injection form TQB3142 in patients with advanced solid tumors.
Peak concentration Cmax | Up to 4 month
  After a single dose, the highest point of the drug-time curve is called the peak concentration.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital , College of Medicine, Zhejiang University, Hangzhou, Zhejiang